CLINICAL TRIAL: NCT00709059
Title: A Non-interventional Phase IV Survey to Assess the Antiviral Effectiveness of PegIntron® and Rebetol® Treatment According to the Stage of Liver Fibrosis in Previously Untreated Patients With Genotype 1/4/5/6 Chronic Hepatitis C (CHC) (PRACTICE)
Brief Title: Efficacy of PegIntron and Rebetol in Previously Untreated Patients With Chronic Hepatitis C Infected With HCV Genotype 1/4/5/6 (Study P04243)
Acronym: PRACTICE
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04243
Record Dates: First submitted 2008-06-23; First posted 2008-07-03 (Estimated); Results first posted 2011-01-10 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PegIntron Plus Rebetol: Previously untreated patients infected with HCV genotype 1, 4, 5, or 6.
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: Rebetol (ribavirin; SCH 18908)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) — PegIntron 1.5 ug/kg body weight per week subcutaneously for 48 weeks
  Other Names: SCH 54031
Drug: Rebetol (ribavirin; SCH 18908) — Rebetol administered based on body weight 800-1200 mg/day (<65 kg: 800 mg; 65 - 85 kg: 1000 mg; >85 kg: 1200 mg) orally for 48 weeks
  Other Names: SCH 18908

SUMMARY:
The objective of the study is to evaluate the effectiveness of PegIntron plus Rebetol combination in treating patients with chronic hepatitis C in a primary care setting. Patients received no antiviral therapy prior to the current study. Only patients infected with Hepatitis C Virus (HCV) genotype 1, 4, 5, or 6 will be enrolled in the study. The study will also explore the influence of liver fibrosis stage on the chances of achieving a sustained virologic response.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated ('treatment naïve') adults (18 year or more) for whom the treating physician has decided to start treatment with PegIntron and Rebetol
* Detectable Hepatitis C Virus - Ribonucleic Acid (HCV-RNA) in serum by Polymerase Chain Reaction (PCR)
* Repeated (with at least a 1 month interval) serum transaminase (alanine aminotransferase [ALT]) levels above the upper normal limit for gender
* Documented chronic hepatitis C (CHC) of genotype 1/4/5/6
* A representative liver biopsy within 1 year prior to inclusion, allowing fibrosis grading into METAVIR score F0, F1, F2, F3 or F4

Exclusion Criteria:

* Known hypersensitivity for any active ingredient or constituent
* Pregnancy or lactation
* Medically documented history of severe psychiatric disturbance, including severe depression, suicidal ideation or suicide attempt
* Medically documented history of severe heart disease, including unstable or uncontrolled cardiac disease, within the last 6 months
* Severely weakening medical condition, including chronic renal insufficiency or creatinine clearance <50 mL/minute
* Hepatitis of immunologic origin or medically documented history of auto-immune disease
* Severe hepatic disorder or decompensated cirrhosis
* Pre-existing thyroid disorder, except if under control with classical treatment
* Epilepsy or central nervous system disorder
* Hemoglobin pathology, eg, thalassaemia, sickle cell anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously untreated patients with chronic hepatitis C, infected with HCV genotype 1, 4, 5, or 6, receiving treatment with PegIntron and Rebetol.
Sampling Method: Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2004-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- PegIntron Plus Rebetol: Previously untreated patients infected with Hepatitis C Virus (HCV) genotype 1, 4, 5, or 6.
Period: Overall Study
Arm/Group | PegIntron Plus Rebetol
Started | 538
Completed | 444
Not Completed | 94
Not completed — Lost to Follow-up | 34
Not completed — Withdrawal by Subject | 19
Not completed — Physician Decision | 7
Not completed — Disease complication | 3
Not completed — Side effects | 20
Not completed — Serious side effects | 11

BASELINE CHARACTERISTICS:
Arm/Group | PegIntron Plus Rebetol
Number analyzed (Participants) | 538
Age, Customized [Number; unit: Participants]
  <50 years | 301
  >=50 years | 204
  age not available | 33
Sex/Gender, Customized [Number; unit: Participants]
  Female | 203
  Male | 302
  Gender not available | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants Who Had a Virological Response (VR) at Week-72
Description: VR was defined as the absence of Hepatitis C virus Ribonucleic Acid (HCV RNA) in a qualitative Polymerase Chain Reaction (PCR) test.
  Participants who dropped out or were withdrawn from treatment were considered not to respond.
Time Frame: Treatment Week 72
Population: Full Analysis Set (FAS)was analyzed. FAS consisted of all participants in the intent-to-treat population wih non-missing viral response at Week 72.
Measure: Number; unit: Participants
Arm/Group | PegIntron Plus Rebetol
Number analyzed (Participants) | 505
Participants | 176

ADVERSE EVENTS:
Description: Per protocol, non-serious adverse events and serious adverse events were not required to be captured as part of the study database.
Arm/Group | PegIntron Plus Rebetol
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The participating physician (PP) agrees not to publish/present any

interim results of the Survey without prior written consent of Schering-

Plough (SP). The PP further agrees to provide 30 days written notice to SP prior to submission for publication or presentation to permit SP to review and comment on any presentation, which right shall include editorial rights. If the parties disagree, the PP agrees to meet with SP to discuss and resolve any such issues or disagreement.